CLINICAL TRIAL: NCT05993013
Title: Improving Strength and Balance in Older Adults at Risk of Falls With the LudoFit Exercise Program
Brief Title: Improving Strength and Balance Through Exercise With LudoFit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Huang (Other)
Collaborators: Jintronix (Unknown)
Responsible Party: Sponsor-Investigator, Shirley Huang, Clinical Investigator, Ottawa Hospital Research Institute
Organization: Ottawa Hospital Research Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4829
Record Dates: First submitted 2023-07-20; First posted 2023-08-15 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Accidental Falls
Keywords: Geriatric medicine; Falls risk; Exercise; Technology
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional exercise (No Intervention): Normally physiotherapist-recommended, tailored strength and balance exercises. These exercises are given in printed handouts and demonstrated by our physiotherapist with the patients during their initial clinic visit. Exercise is recommended to be done at least 3 times per week.
- Game-based exercise (Experimental): Strength and balance exercises using the LudoFit game-based exercise software. Participants will be registered on the platform. Exercise is recommended to be done at least 3 times per week.
  Interventions: Other: LudoFit

INTERVENTIONS:
Other: LudoFit — Game-based, technology-enabled home exercise software, done at least 3 times per week. Video games for a variety of exercises that promote balance, strength, endurance, and coordination.
  Arms: Game-based exercise

SUMMARY:
The goal of this mixed methods cohort study is to explore how an innovative game-based, technology-enabled home exercise software compares to a conventional home-based exercise program in older adults at risk for falls. The main question[s] it aims to answer are:

* Does the exercise software lead to better or similar adherence to exercise recommendations compared to the conventional exercise program?
* Does the exercise software improve user strength and balance, as measured by relevant physical function scores?
* Do participants find the exercise software enjoyable and acceptable?

Participants will be approached during their initial fall risk assessment to see if they are interested in taking part. Those who agree to participate will choose either the exercise software or the conventional exercise program and will be instructed to:

* Perform their respective exercise program for a minimum of 3 times a week for 3 months.
* Return to clinic in 3 months to see our C-FAST physiotherapist for reassessment of their relevant physical functional tests.
* For conventional exercise program only - Document exercise compliance in an exercise log.
* For software program only - Complete a survey regarding the use of the technology.

Researchers will compare software-use cohort versus conventional exercise program cohort to see if adherence and physical function scores are comparable.

DETAILED DESCRIPTION:
This study will take place in the Champlain Falls Assessment and Streamlined Treatment (C-FAST) clinic at the Ottawa Hospital, Division of Geriatric Medicine. This clinic receives patient referrals from the community for fall risk assessment. It strives to see older adults early in their 'falls history' with the goal of promoting their independence and avoiding unnecessary health care utilization due to falls and related injuries. Each patient receives a comprehensive fall risk assessment and individualized, evidenced-based, interventions/recommendations to address their fall risk, including physiotherapist-prescribed strength and balance exercises. The investigators want to find out whether delivering a home-based exercise program using video game-based technology may be acceptable to our patient population and possibly improve adherence to exercise intervention. The investigators will partner with Jintronix, a company that was founded to bring interactive technology to rehabilitation and senior care. LudoFit is one of Jintronix' s latest software programs where older adults participate in strength and balance exercises using an innovative game-based, technology-enabled home exercise software. The investigators want to conduct a study in our clinic where older adults have the option of choosing to exercise using LudoFit software instead of the conventional home-based exercise program and to see whether they show good compliance to exercises, improvement in their specific strength and balance scores and find this method an acceptable and fun way to exercise.

ELIGIBILITY:
Inclusion Criteria:

* Patient is interested in a home-based exercise program.
* The patient is independent with activities of daily living and instrumental activities of daily living.
* Patient agrees to return for 3-month follow-up.
* Patient must speak English or French.

Exclusion Criteria:

* Patient has the following physical functional performance:

  1. Berg Balance Scale score of 45 or less
  2. Unable to safely and independently reach at least 5 inches to the side and forward
  3. Unable to safely and independently reach down, touch floor and then return to start position
* Patient has diagnosed or suspected cognitive impairment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Physical function test 1-Berg Balance Scale | 3 months
  Berg Balance Scale is a series of balance maneuvers administered by a physiotherapist to assess the balance of a subject. It is scored from 0 to 56. The higher the score the better the balance. Subject scores are also compared to age-matched normative values. This measure will be collected at initial clinic visit and then again at 3-month follow-up visit and the values compared for any improvement.
Physical function test 2-Timed Up and Go Test | 3 months
  Timed Up and Go Test documents time taken in seconds for a subject stand up from a chair, walk 3 meters forward and then return to the chair and sit down. The longer the time taken, the worse the outcome. Taking over 14 seconds in Timed Up and Go Test correlates with increased risk of falls. This measure will be collected at initial clinic visit and then again at 3-month follow-up visit and the values compared for any improvement.
Physical function test 3-Five Time Sit to Stand Test | 3 months
  Five Times Sit to Stand test scoring is based on the amount of time (to the nearest decimal in seconds) a subject is able to transfer from a seated to a standing position and back to sitting five times. The lower the time to complete the test the better the outcome of the test. Subject scores are also compared to age-matched normative values. This measure will be collected at initial clinic visit and then again at 3-month follow-up visit and the values compared for any improvement.
Conventional exercise cohort - Exercise adherence | 3 months
  Participants will be given an exercise log at the beginning of the study and asked to use this log to document frequency of exercise each week, minutes spent during each exercise session and any additional comments/feedback about each exercise session (e.g. any discomfort or difficulty performing the exercise). The researchers will collect the exercise log at the 3-month follow-up visit and the entries analyzed. The more frequently the exercises were performed measured in total number of days per week and total minutes spent exercising, the better. Any qualitative comments provide by subjects in the log will be collected and analyzed for any themes.
LudoFit exercise cohort - Exercise adherence | 3 months
  LudoFit software automatically tracks user exercise adherence data, including minutes of use per day, as well as performance in each activity and rate of perceived exertion. This data will be downloaded by researchers and analyzed. The more frequently the exercises were performed measured in total number of days per week and total minutes spent exercising, the better.

SECONDARY OUTCOMES:
Satisfaction with LudoFit exercise software | 3 months
  Participants will be given a standardized paper survey to complete at the 3-month follow-up visit where they will answer questions pertaining to their user experience with the software, such as acceptability and usability. The survey includes both quantitative (13 statements where subjects rate their agreement with the statements on a 5-point Likert scale; the higher the score, the higher the agreement with the statement) and qualitative components (subjects can provide additional comments to express what they find most beneficial with using LudoFit software and what could have made their experience with LudoFit better).

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada